CLINICAL TRIAL: NCT01444404
Title: A Phase 1, First-In-Human Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacokinetics of AMG 820 in Adult Subjects With Advanced Solid Tumors
Brief Title: A Study of AMG 820 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AmMax Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20060347
Record Dates: First submitted 2011-09-01; First posted 2011-09-30 (Estimated); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Advanced Malignancy; Advanced Solid Tumors; Cancer; Oncology; Oncology Patients; Tumors
Keywords: Solid Tumors; Phase 1; Clinical Trial
MeSH Terms: conditions — Neoplasms

ARMS (2):
- Dose Expansion (Experimental): The dose expansion will consist of up to 20 subjects and the dose level of AMG 820 will be dependent upon emerging safety and PK data from the dose escalation part of the study.
  Interventions: Drug: AMG 820
- Dose Escalation (Experimental): The dose escalation part of the study is aimed at evaluating the safety, tolerability, pharmacokinetics and pharmacodynamics of AMG 820.
  Interventions: Drug: AMG 820

INTERVENTIONS:
Drug: AMG 820 — AMG 820 is a fully human IgG2 c-fms antagonistic antibody and will be given every two weeks until progression or unacceptable toxicity develops.

SUMMARY:
First in human, open-label, sequential dose escalation and expansion study of AMG 820 in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 years old
* Subjects must have a pathologically documented, definitively diagnosed, advanced solid tumor
* Measurable disease per RECIST 1.1 guidelines
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
* Part 2 - Dose Expansion only: Subjects must have tumor tissue that is accessible for core needle biopsy by using minimally invasive procedures and must consent to undergo biopsies of the tumor
* Able to fast 4 to 6 hours for FDG-PET/CT scan, except subjects with prostate or bladder cancers
* Competent to sign and date an Institutional Review Board approved informed consent form
* Adequate hematologic, renal and hepatic function as determined by laboratory blood and urine tests

Exclusion Criteria:

* Men and woman of reproductive potential, unwilling to practice a highly effective method of birth control for the duration of the study and an additional 4 months after receiving the last dose of study drug.
* Women who are lactating/breastfeeding or planning to become pregnant during the duration of the study
* Primary central nervous system (CNS) tumors or CNS metastases
* History of presence of hematological malignancies
* History of arterial or venous thrombosis within 6 months of study enrollment
* History of bleeding diathesis
* Myocardial infarction within 6 months of study day 1, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or unstable cardiac arrhythmia requiring medication, or uncontrolled hypertension
* Hypertension not adequately controlled with medication (diastolic > 90mmHG; systolic > 140 mmHG)
* Left ventricular ejection fraction (LVEF) ≤ 50%
* Active infection requiring (IV) antibiotics within 2 weeks of study enrollment
* Known positive test for human immunodeficiency virus (HIV)
* Known chronic hepatitis B or hepatitis C infection
* Positive test for hepatitis B surface antigen or hepatitis C antibody
* Known history of tuberculosis (TB), exposure to active TB-infected individuals, or positive TB skin test (tuberculin or purified protein derivative (PPD) test) upon study entry (subjects previously vaccinated for TB are not excluded unless there is evidence of active TB)
* Anti-tumor therapy within 4 weeks of study day 1 including chemotherapy, antibody therapy, retinoid therapy, or other investigational agent
* Concurrent or prior anticoagulation therapy within 28 days of study day 1
* Major surgery within 28 days of study day 1
* Any co-morbid medical disorder that may increase the risk of toxicity, in the opinion of the investigator or sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-03-31 (Actual); Primary Completion 2014-02-06 (Actual); Study Completion 2014-02-06 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) Time Frame: predose, 0.5, 1, 2, 4, 8, 24 hours post-dose | 3 years
Dose of AMG 820 where clinically significant or ≥ Grade 3 changes in safety laboratory tests, physical examinations, ECGs, or vitals signs in all subjects enrolled is greater than 33%. | 3 years
Change in tumor associated macrophages (TAMS) as assessed by tumor biopsy at 9 weeks. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, San Antonio, Texas

REFERENCES:
- [Background] Papadopoulos KP, Gluck L, Martin LP, Olszanski AJ, Tolcher AW, Ngarmchamnanrith G, Rasmussen E, Amore BM, Nagorsen D, Hill JS, Stephenson J Jr. First-in-Human Study of AMG 820, a Monoclonal Anti-Colony-Stimulating Factor 1 Receptor Antibody, in Patients with Advanced Solid Tumors. Clin Cancer Res. 2017 Oct 1;23(19):5703-5710. doi: 10.1158/1078-0432.CCR-16-3261. Epub 2017 Jun 27. PMID 28655795
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com